CLINICAL TRIAL: NCT02617355
Title: Interference Between Surgical Magnetic Drapes and Pacemakers: An Observational Study Comparing Commercially Available Devices and a New Magnetically Isolated Drape
Brief Title: Interference Between Surgical Magnetic Drapes and Pacemakers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Valerie Zaphiratos, Clinical associate Professor, Maisonneuve-Rosemont Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11061
Record Dates: First submitted 2015-11-24; First posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Electromagnetic Interference

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prototype vs Covidien magnetic drape (Other): New prototype surgical magnetic drape made with bottom-isolated ferrite magnets applied to the patient's thorax vs Covidien magnetic drape
  Interventions: Device: Prototype surgical magnetic drape; Device: Green Covidien Magnetic Drape
- Prototype vs 4 commercial drapes (Other): New prototype surgical magnetic drape made with bottom-isolated ferrite magnets applied to the patient's thorax vs 4 commercially available magnetic drapes:
  Green Covidien Magnetic Drape Jac-Cell Medic Reusable Magnetic Pad DeRoyal Magnetic Pad size 10" x 16" DeRoyal Magnetic Pad size 20" x 16"
  Interventions: Device: Prototype surgical magnetic drape; Device: Green Covidien Magnetic Drape; Device: Jac-Cell Medic Reusable Magnetic Pad; Device: DeRoyal Magnetic Pad size 20" x 16"; Device: DeRoyal Magnetic Pad size 10" x 16"

INTERVENTIONS:
Device: Prototype surgical magnetic drape — New prototype surgical magnetic drape made with bottom-isolated ferrite magnets applied to the patient's thorax
Device: Green Covidien Magnetic Drape — Green Covidien Magnetic Drape applied to the patient's thorax
Device: Jac-Cell Medic Reusable Magnetic Pad — Jaa-Cell Medic Reusable Magnetic Pad applied to the patient's thorax
  Arms: Prototype vs 4 commercial drapes
Device: DeRoyal Magnetic Pad size 20" x 16" — Magnetic Instrument Pad #25-002, size 20" x 16", DeRoyal Industries Inc applied to the patient's thorax
  Arms: Prototype vs 4 commercial drapes
Device: DeRoyal Magnetic Pad size 10" x 16" — Magnetic Instrument Pad #25-001, size 10" x 16", DeRoyal Industries Inc applied to the patient's thorax
  Arms: Prototype vs 4 commercial drapes

SUMMARY:
This study is designed to compare a new prototype surgical magnetic drape made with bottom-isolated ferrite magnets to 4 commercially available surgical magnetic drapes.

DETAILED DESCRIPTION:
Magnetic fields may potentially interfere with the function of cardiovascular implantable electronic devices. Sterile magnetic drapes used to hold surgical instruments are often placed on the patient's thorax, and they are likely to interfere with the function of these devices.

This study compares the magnetic interference of a new prototype surgical magnetic drape made with bottom-isolated ferrite magnets to the Covidien magnetic drape and 3 other commercially available surgical magnetic drapes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pacemaker
* 18 years or older

Exclusion Criteria:

* Patients with implantable cardioverter-defibrillator (ICD)
* Patients in whom the magnet rate cardiac rhythm is indistinguishable from their baseline rhythm
* Refusal/Inability to consent
* Language other than French or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Percentage of magnetic interference | Within 2 minutes after placement of surgical magnetic drape to the patient's chest
  Percentage of patients experiencing magnetic interference with the application of each surgical magnetic drape.
  Magnetic interference defined as a cardiac rhythm change to asynchronous and identical to that produced by a round magnet rhythm over the pacemaker.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Zaphiratos, MD, Principal Investigator — Maisonneuve-Rosemont Hospital